CLINICAL TRIAL: NCT06619847
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study Evaluating the Efficacy and Safety of VX-993 for Acute Pain After a Bunionectomy
Brief Title: A Study Evaluating Efficacy and Safety of VX-993 for Acute Pain After a Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-993-101
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VX-993 (Experimental): Participants will be randomized to receive different dose levels of VX-993.
  Interventions: Drug: VX-993; Drug: Placebo (matched to HB/APAP)
- Hydrocodone bitartrate/acetaminophen (HB/APAP) (Active Comparator): Participants will be randomized to receive HB/APAP.
  Interventions: Drug: HB/APAP; Drug: Placebo (matched to VX-993)
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-993 and HB/APAP.
  Interventions: Drug: Placebo (matched to VX-993); Drug: Placebo (matched to HB/APAP)

INTERVENTIONS:
Drug: VX-993 — Tablets for oral administration.
  Arms: VX-993
Drug: HB/APAP — Capsules for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP)
Drug: Placebo (matched to VX-993) — Placebo matched to VX-993 for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP); Placebo
Drug: Placebo (matched to HB/APAP) — Placebo matched to HB/APAP for oral administration.
  Arms: Placebo; VX-993

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of VX-993 in treating acute pain after a bunionectomy.

ELIGIBILITY:
Key Inclusion Criteria:

Before Surgery:

* Participant scheduled to undergo a primary unilateral bunionectomy with distal first metatarsal osteotomy (i.e., Austin procedure) and internal fixation under regional anesthesia (Mayo block)

After Surgery:

* Participant is lucid and able to follow commands
* All analgesic guidelines were followed during and after the bunionectomy

Key Exclusion Criteria:

Before Surgery:

* Prior history of bunionectomy or other foot surgery on the index foot
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s) within the last 2 years
* A known or clinically suspected active infection with human immunodeficiency virus or hepatitis B or C viruses

After Surgery:

* Participant had a Type 3 deformity requiring a base wedge osteotomy or concomitant surgery such as hammertoe repair, or had medical complications during the bunionectomy

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference (SPID) as Recorded on the Numeric Pain Rating Scale (NPRS) From 0 to 48 Hours (SPID48) | From 0 to 48 Hours After the First Dose of Study Drug

SECONDARY OUTCOMES:
Proportion of Participants With Greater Than or Equal To (>=) 30 Percent (%) Reduction in NPRS at 48 Hours | At 48 Hours After the First Dose of Study Drug
Proportion of Participants With >=50% Reduction in NPRS at 48 Hours | At 48 Hours After the First Dose of Study Drug
Proportion of Participants With >=70% Reduction in NPRS at 48 Hours | At 48 Hours After the First Dose of Study Drug
Maximum Observed Plasma Concentration (Cmax) of VX-993 and its Metabolite | Pre-dose to 12 Hours and 24 to 36 Hours After the First Dose of Study Drug
Area Under the Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-993 and its Metabolite | Pre-dose to 12 Hours and 24 to 36 Hours After the First Dose of Study Drug
Time to Reach Maximum Observed Plasma Concentration (Tmax) of VX-993 and its Metabolite | Pre-dose to 12 Hours and 24 to 36 Hours After the First Dose of Study Drug
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 19

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Shoals Medical Trials Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Trovare Clinical Research, Bakersfield, California
  - New Hope Research Development | Tarzana, CA, Tarzana, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - BioBehavioral Research of Austin, Austin, Texas
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - HD Research LLC | Legent Orthopedic Hospital, Carrollton, Texas
  - Memorial Hermann Village, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing